CLINICAL TRIAL: NCT04802421
Title: Hemodynamic Effect of Alveolar Recruitment Manoeuver Through Stepwise Increase and Decrease in Irway Pressure or Sustained 30 Secondes 30 cmH2O Continuous Positive Airway Pressure. A Randomized Study.
Brief Title: Effect Alveolar Recruitment Manoeuver on Stroke Volume a Randomized Study
Acronym: hemorecrut-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CHU Caen Normandie 19-024
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Alveolar Recruitment Manoeuver; Anesthesia

STUDY DESIGN:
Intervention Model Description: randomised parallel groups. randomisation between 2 groups equilibated by randomised blocks of 4, 6 or 8
Who Masked: Participant, Care Provider
Masking Description: The patient will not know the allocation group because he will be anesthetised before randomisation. The care provider (anesthetist) will not know the allocation group because the intervention will be applied by an independent investigator not involved in care of the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP30 (Active Comparator): a 30 secondes 30 cmH2O continuous positive airway pressure applied after the orotracheal intubation will be checked and secured following induction of general anesthesia
  Interventions: Procedure: alveolar recruitment manoeuver
- STEP30 (Active Comparator): a stepwise increase (+5 cmH2O) in postivie airway pressure from +5 cmH2O to +30 cmH2O and decrease (-5 cmH2O) from +30 cmH2O to +5 cmH2O applied after the orotracheal intubation will be checked and secured following induction of general anesthesia
  Interventions: Procedure: alveolar recruitment manoeuver

INTERVENTIONS:
Procedure: alveolar recruitment manoeuver — alveolar recruitment manoeuver are recommended during general anesthesia to prevent pulmonary atelectasis

SUMMARY:
Objective: to compare the effect of alveolar recruitment manouver through stepwise increase and decrease in airway pressure or sustained 30 secondes 30 cmH2O continuous positive airway pressure on cardiac stroke volume estimated by oesophageal doppler in preload independent anesthetized patients scheduled for surgery.

DETAILED DESCRIPTION:
Following anesthesia and preload optimisation guided by cardiac stroke volume, patients will be randomised to one alveolr recruitment manoeuver :

* stepwise increase and decrease in positive airway pressure
* sustained 30 secondes 30 cmH2O continuous positive airway pressure The primary objective is the change in cardiac stroke volume.

ELIGIBILITY:
Inclusion Criteria:

* adult patients scheduled for major surgery requiring hemodynamic monitoring
* written signed informed consent

Exclusion Criteria:

* pregnancy
* non sinusal heart rate
* known cardiac right ventricular failure or arterial pulmonary hypertension
* pneumothorax
* known pulmonary emphysema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
cardiac stroke volume | 1 min
  change in cardiac stroke volume during the alveolar recruitment manoeuver

SECONDARY OUTCOMES:
arterial pressure | 1 min
  change in arterial pressure during the alveolar recruitment manoeuver
recovery at 3 min | 3 min
  recovery of cardiacstroke volume and arterial pressure 3 min after the end of alveolar recruitment manoeuver

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Caen, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dupont K, Lefrancois V, Delahaye A, Sanz M, Hestin R, Doublet T, Parienti JJ, Hanouz JL. Change in stroke volume during alveolar recruitment maneuvers through transient continuous positive airway pressure or stepwise increase in positive end expiratory pressure in anesthetized patients: a prospective randomized double-blind study. Can J Anaesth. 2024 Feb;71(2):224-233. doi: 10.1007/s12630-023-02644-7. Epub 2023 Nov 28. PMID 38017197